CLINICAL TRIAL: NCT03539965
Title: Triple-negative Breast Cancer: a New Perspective on Predictive and Prognostic Biomarkers
Brief Title: Triple-negative Breast Cancer: a New Perspective on Biomarkers
Acronym: TNBCbrazil
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Jesse Lopes da Silva, MD, Instituto Nacional de Cancer, Brazil
Other Study IDs: TNBCbrazil
Record Dates: First submitted 2018-05-04; First posted 2018-05-30 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Triple Negative Breast Neoplasms; Triple Negative Breast Cancer
Keywords: Neoadjuvant Chemotherapy; Predictive Biomarkers; Prognostic Biomarkers; Complete Pathological Response; Tumor Infiltrating Lymphocytes; PD-L1; PD-L2
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Paraffin-embedded Hematoxylin & Eosin (H & E) core biopsy/early biopsy and surgical specimens previously analyzed in the Department of Patology of the Brazilian National Cancer Institute (INCA) will be doubly reviewed by two pathologists in our study for histological grade (Scarff-Bloom-Richardson method, modified by Elston and Ellis), histological type (according to World Health Organization, 2012), presence of carcinoma component "in situ", angiolymphatic invasion, perineural infiltration, presence of lymphocytic inflammatory infiltrate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-arm cohort: Initially, patients will be analyzed in a single group. After determining the status of the biomarkers, the patient sample will be divided into specific groups for comparative purposes.

SUMMARY:
A single-institutional cohort to determine the prevalence of new immunohistochemical panel in advanced triple-negative submitted to neoadjuvant chemotherapy and its association with response and survival.

DETAILED DESCRIPTION:
Background/Rationale: Triple negative breast cancer (TNBC) is known to be a heterogeneous disease, and different molecular sub-classifications are proposed based in specific biomarkers as immunohistochemical (IHC) expression of the androgen-receptor (AR), Epidermal growth Factor Receptor (EGFR), Cytokeratin 5/6 (CK5/6), Cytokeratin14 (CK14), Cytokeratin 17 (CK17), clusters of differentiation 117 (CD 117), p53, Ki67 level, Programmed cell death-ligand 1 (PD-L1) and PD-L2 in tumor cell membrane and the pattern of tumor infiltrating mono-lymphocytes (PD-1+, FOXP3+, CD 4+ or cluster designation 8 (CD8 +), CD 3+, cluster of differentiation 56 (CD56+), cluster designation 68 (CD68+) or CD 14+). Predicting response and survival to neoadjuvant treatment of locally advanced triple-negative breast cancer remains a major challenge. Many doubts still prevail over the role of new biomarkers in predicting different outcomes for tumors with the same stage and morphological characteristics.

Objectives and Hypotheses:

Primary objective: To evaluate the association of the intratumoral lymphocytic infiltrate (TILs) status profile in the core biopsy with complete pathological response (CPR) outcomes to neoadjuvant chemotherapy and progression-free survival (PFS). Secondary objectives: To evaluate the association of the others biomarkers expression profile and the quality of TILs with PFS and CPR. To determine the prevalence of a large immunohistochemical panel (AR, EGFR, CK5/6, CK14, CK17, CD 117, p53, Ki67 level, PD-L1 and PD-L2 in tumor cell membrane and the pattern of tumor infiltrating mono-lymphocytes PD-1+, FOXP3+, CD 4+ , CD8 +, CD 3+, CD56+, CD68+ and/or CD 14+), before and after neoadjuvant chemotherapy. To determine if the negativation of biomarkers after the systemic treatment is associated with CPR and PFS.

Methods:

Study design: A cohort with retrospective data collection and sectional analysis of pathological material.

Data Source(s): Medical records and pathological material. Study Population: Women with locally advanced triple negative breast cancer consecutively enrolled at Brazilian National Cancer Institute (INCA) submitted to neoadjuvant treatment and subsequently operated.

Exposure(s): Status of specified biomarkers. Outcome(s): Complete Pathologic Response and Progression free Survival and Sample Size Estimations: With a type I error of 5% and study power of 80%, it is estimated that 155 patients are needed.

Statistical Analysis: Statistical analysis will be performed using SPSS (version 18.0 for windows, statistical package for social science (SPSS) Inc., Chicago, IL). Survival curves will be constructed using the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years
* Locally advanced TNBC (T3-4, any Node, M0; any Tumor, N1-3, M0)
* Patients submitted to anthracycline and taxane-based neoadjuvant chemotherapy and then operated between January 2010 and December 2014 at the Brazilian National Cancer Institute.

Exclusion Criteria:

* Patients with metastatic Breast Cancer;
* Other non-epithelial histologies of breast cancer;
* Pure Ductal Carcinoma In Situ diagnoses are not eligible.
* Patients with scarce material for immunohistochemistry;
* Other primary synchronous or anachronistic tumors in the breast or other sites;
* No prior immunotherapeutic, chemotherapeutic or antiandrogenic drugs allowed
* Patients treated with alternative neoadjuvant chemotherapy regimens (not based on anthracycline and taxane) or with only hormone therapy;
* Patients who received chemotherapy or who were operated outside the INCA.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who is biopsied and diagnosed with breast cancer in the public health system is referred to Brazilian National Cancer Institute (INCA) through a registry and screening performed by the Municipal Health Department of the city of Rio de Janeiro. Therefore, it becomes a great field for research of cancer patients by the large number of cases. Absolutely all patients enrolled in INCA for treatment have their biopsy material reviewed in DIPAT.
  In this cohort, will be studied women with locally advanced TNBC consecutively enrolled at INCA between January 2010 and December 2014 that were submitted to neoadjuvant chemotherapy and subsequently operated.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Approximately 24 months: from diagnosis up to the first event defined as local recurrence or distant relapse, or death, whichever come first through study completion.
  The first event defined as local recurrence or distant relapse, or death, whichever come first.

SECONDARY OUTCOMES:
Clinical Response Rate | From date of first cycle of chemotherapy until completion of neoadjuvant treatment, approximately 16 weeks
  To determine the clinical response rate in patients with palpable disease.
Objective response rate | From date of first cycle of chemotherapy until completion of neoadjuvant treatment, approximately 16 weeks
  To compare overall objective response rate in both treatment groups.
Determine predictive markers | Approximately 24 weeks: from diagnosis up to surgery.
  To determine predictive markers for sensitivity and resistance to chemotherapy.
Determine prognostic markers | Approximately 24 months: from diagnosis up to the first event defined as local recurrence or distant relapse, or death, whichever come first through study completion.
  To determine prognostic markers for progression free survival after neoadjuvant chemotherapy and surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse L da Silva, MD, Principal Investigator — Instituto Nacional de Cancer
Locations (1):
- Instituto Nacional do Cancer - CPQ, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No